CLINICAL TRIAL: NCT02986048
Title: Proton Therapy Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE4Y16
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Treatment With Proton Beam Radiation Therapy
Keywords: proton beam; registry; radiation; cancer
MeSH Terms: conditions — Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proton Beam Therapy: All patients treated with proton beam therapy at the UH Proton Therapy Center who consent to have their health information recorded, including whether the cancer was cured and if any complications occur ed due to treatment
  Interventions: Other: Proton Beam Therapy

INTERVENTIONS:
Other: Proton Beam Therapy — Intervention is not assigned. Only patient data is being collected

SUMMARY:
The purpose of this study is to establish a database (or "registry") of patients treated with proton beam therapy at the University Hospitals (UH) Proton Therapy Center. By keeping track of the patients treated it will allow the investigators to periodically evaluate the outcomes of patients.

DETAILED DESCRIPTION:
The primary objective of this non-therapeutic registry study is to create a secure longitudinal database of patients treated with proton therapy at the UH Proton Therapy Center. This will allow reporting patient, tumor, and treatment characteristics as well as outcome data pertaining to disease control and complications for this relatively rare radiation modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with proton beam at the UH Proton Therapy Center
* Patients who have the ability to understand and be willing to sign a written informed consent document

Exclusion Criteria:

* Patients or legal guardians who are unable to understand informed consent document

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with proton beam at the UH Proton Therapy Center
Sampling Method: Non-Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2016-11-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants treated at UH Proton Therapy Center by proton beam therapy | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: David B Mansur, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States